## **Study Protocol Cover Sheet**

| Official Title: |
|---|
| A Comparative Evaluation of Quadratus Lumborum Block Versus Fascia Iliaca Nerve |
| Block for Patients Undergoing Elective Total Hip Replacement Under Spinal Anaesthesia |
| NCT number: |
| not yet known |
| Unique Protocol ID: |
| 2017/1/01-2018-01 |
| Date of document: |
| 30/04/2018 |

## **CONSENT FORM**

Title of Research Study: A COMPARATIVE EVALUATION OF QUADRATUS LUMBORUM BLOCK VERSUS FASCIA ILIACA NERVE BLOCK FOR PATIENTS UNDERGOING ELECTIVE TOTAL HIP REPLACEMENT UNDER SPINAL ANAESTHESIA

| Patient Details | |
|-----------------|-----|
| Name | MRN |
| D.O.B | |
| Add | |
| M/F | |

This study and this consent form have been explained to me. My doctor has answered all my questions to my satisfaction. I believe I understand what will happen if I agree to be part of this study. I have read, or had read to me, this consent form. I have had the opportunity to ask questions and all my questions have been answered to my satisfaction. I freely and voluntarily agree to be part of this research study, though without prejudice to my legal and ethical rights. I agree to the following

- Randomisation
- Block procedure
- Pre and post block test related to the study
- Use of data

I have received a copy of this agreement.

| PARTICIPANT'S NAME: | |
|-------------------------------------------------------------------|---|
| PARTICIPANT'S SIGNATURE: | _ |
| Date: | |
| Date on which the participant was first furnished with this form: | |
| NAME OF CONSENTOR, PARENT or GUARDIAN: | |
| SIGNATURE: | |
| RELATION TO PARTICIPANT: | |

Where the participant is capable of comprehending the nature, significance and scope of the consent required, but is physically unable to sign written consent, signatures of two witnesses present when consent was given by the participant to a registered medical practitioner treating him or her for the illness.

| NAME OF FIRST | WITNESS: |
|---------------|----------|

| SIGNATURE: |
|---|
| NAME OF SECOND WITNESS: |
| SIGNATURE: |
| Statement of investigator's responsibility: |
| I have explained the nature, purpose, procedures, benefits, risks of, or alternatives to, this |
| research study. I have offered to answer any questions and fully answered such questions. |
| believe that the participant understands my explanation and has freely given informed |
| consent. |
| Physician's signature: |
| Date: |

(Keep the original of this form in the participant's medical record, give one copy to the participant, keep one copy in the investigator's records, and send one copy to the sponsor (if there is a sponsor).